CLINICAL TRIAL: NCT03563781
Title: SEntine Lymph Node in earLY Ovarian Cancer
Brief Title: SEntine Lymph Node in earLY Ovarian Cancer (SELLY)
Acronym: SELLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SCAMBIA GIOVANNI, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CICOG-2-3-18/12
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Sentinel Lymph Node; Ovarian Cancer Stage I
Keywords: ovarian cancer; laparoscopy; sentinel node; lymphadenectomy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients with early ovarian cancer will receive sentinel node procedure before full lymphadenectomy, in order to assess the accuracy of sentinel node in diagnosing the presence of nodal metastases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SENTINEL NODE (Other): Patients with ovarian cancer will receive sentinel node identification and they will be then submitted to complete pelvic and para-aortic lymphadenectomy (as per the present guidelines)
  Interventions: Procedure: Sentinel node detection

INTERVENTIONS:
Procedure: Sentinel node detection — Patients will receive injection of tracer in the ovarian ligaments to identify the lymphatic drainage of the affected ovary and ultimately the sentinel node. Afterwards, systematic lymphadenectomy will be accomplished according to current guidelines.

SUMMARY:
The present study aims at investigating the feasibility, the detection rate and the negative predictive value of sentinel node in predicting the presence or absence of lymph node metastasis in ovarian cancer patients

DETAILED DESCRIPTION:
Patients with early stage ovarian cancer have a good prognosis. However, nearly 15% of the initially diagnosed as early stage ovarian cancers, will be upstaged after an appropriate surgical staging due to lymphatic metastasis, despite of preoperative radiological data. Therefore, complete pelvic and para-aortic lymphadenectomy in these patients represents a crucial procedure. On the other hand, nodal dissection may be associated with threatening intra- and post-operative complications.

If feasible and accurate, the sentinel lymph node procedure could be a modality to avoid unnecessary radical lymphadenectomy without missing important information on nodal status.

With the present study we aim at exploring the role of sentinel node dissection in early ovarian cancer patients.

Patients with ovarian cancer macroscopically limited to the ovary (early ovarian cancer) will receive injection of a tracer (patent blue or indocyanine green) which have already been proven safe and extremely effective in several other gynecologic and non-gynecologic malignancies. Then the retroperitoneal spaces will be opened as for a standard lymphadenectomy procedure and the lymph node marked with the tracer will be identified. After dissection of the sentinel node, lymphadenectomy will be completed according to current guidelines.

Operative data, pathological findings and accuracy of sentinel node in predicting nodal status will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Epithelial ovarian cancer
* Early stage disease limited to the ovary

Exclusion Criteria:

* Evidence of extraovarian disease
* Allergy to the materials used

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a gynecologic study therefore only biologically female patients will be included
Enrollment: 176 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with procedure-related adverse events | 6 months
  The number of patients with procedure-related adverse events as assessed by CTCAE v4.0
Detection rate | 24 months
  The rate of patients in whom the sentinel node is detected

SECONDARY OUTCOMES:
Negative predictive value | 24 months
  The negative predictive value of sentinel node in assessing nodal status

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Giovannni Scambia, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared only with those making official request to the study investigator
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will become available One year after publication, and they will be available for 6 months.
Access Criteria: Direct request to the study PI

REFERENCES:
- [Result] Uccella S, Gisone B, Stevenazzi G, Ghezzi F. Laparoscopic sentinel node detection with ICG for early ovarian cancer: Description of a technique and literature review. Eur J Obstet Gynecol Reprod Biol. 2018 Feb;221:193-194. doi: 10.1016/j.ejogrb.2017.12.004. Epub 2017 Dec 6. No abstract available. PMID 29224846
- [Result] Sadeghi R. Feasibility of Sentinel Node Mapping in Ovarian Tumors: What Is the Evidence? Int J Gynecol Cancer. 2018 Feb;28(2):421-422. doi: 10.1097/IGC.0000000000001158. No abstract available. PMID 29194194
- [Result] Nyberg RH, Korkola P, Maenpaa JU. Sentinel Node and Ovarian Tumors: A Series of 20 Patients. Int J Gynecol Cancer. 2017 May;27(4):684-689. doi: 10.1097/IGC.0000000000000948. PMID 28375928
- [Derived] Scambia G, Nero C, Uccella S, Vizza E, Ghezzi F, Cosentino F, Chiantera V, Fagotti A. Sentinel-node biopsy in early stage ovarian cancer: a prospective multicentre study (SELLY). Int J Gynecol Cancer. 2019 Nov;29(9):1437-1439. doi: 10.1136/ijgc-2019-000886. Epub 2019 Oct 9. PMID 31601646